CLINICAL TRIAL: NCT00499668
Title: A Pilot Study of Aprepitant Versus Ondansetron for the Treatment of Opioid Induced Nausea and Vomiting
Brief Title: Aprepitant or Ondansetron in Treating Nausea and Vomiting Caused By Opioids in Patients With Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: slow accrual
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Barbara Murphy, MD, Professor of Medicine; Director, Cancer Supportive Care Program; Director, Head and Neck Research Program; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VICC SUPP 0513; VU-VICC-SUPP-0513; VU-VICC-IRB-070193; MERCK-VU-VICC-SUPP-0513
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2013-03

CONDITIONS: Myeloproliferative Disorders; Leukemia; Lymphoma; Lymphoproliferative Disorder; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Nausea and Vomiting; Solid Tumor
Keywords: unspecified adult solid tumor, protocol specific; nausea and vomiting; chronic myelogenous leukemia; chronic eosinophilic leukemia; chronic idiopathic myelofibrosis; chronic neutrophilic leukemia; essential thrombocythemia; polycythemia vera; adult acute lymphoblastic leukemia; adult acute myeloid leukemia; acute undifferentiated leukemia; mast cell leukemia; adult T-cell leukemia/lymphoma; T-cell large granular lymphocyte leukemia; chronic lymphocytic leukemia; hairy cell leukemia; prolymphocytic leukemia; AIDS-related lymphoma; adult Hodgkin lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; cutaneous B-cell non-Hodgkin lymphoma; cutaneous T-cell non-Hodgkin lymphoma; mycosis fungoides/Sezary syndrome; adult grade III lymphomatoid granulomatosis; adult nasal type extranodal NK/T-cell lymphoma; Waldenstrom macroglobulinemia; adult Burkitt lymphoma; adult diffuse large cell lymphoma; adult diffuse mixed cell lymphoma; adult diffuse small cleaved cell lymphoma; adult immunoblastic large cell lymphoma; adult lymphoblastic lymphoma; grade 1 follicular lymphoma; grade 2 follicular lymphoma; grade 3 follicular lymphoma; mantle cell lymphoma; marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; small lymphocytic lymphoma; intraocular lymphoma; primary central nervous system lymphoma; post-transplant lymphoproliferative disorder; multiple myeloma and other plasma cell neoplasms; myelodysplastic syndromes; atypical chronic myeloid leukemia; chronic myelomonocytic leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; chronic myeloproliferative disorders; myelodysplastic/myeloproliferative diseases
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Lymphoproliferative Disorders; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Nausea; Vomiting; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Neutrophilic, Chronic; Thrombocythemia, Essential; Polycythemia Vera; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Biphenotypic, Acute; Leukemia, Mast-Cell; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Large Granular Lymphocytic; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Leukemia, Prolymphocytic; Lymphoma, AIDS-Related; Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Extranodal NK-T-Cell; Waldenstrom Macroglobulinemia; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Intraocular Lymphoma; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Myelomonocytic, Chronic; Myelodysplastic-Myeloproliferative Diseases | interventions — Aprepitant; Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARM A (Experimental)
  Interventions: Drug: aprepitant
- ARM B (Experimental)
  Interventions: Drug: ondansetron hydrochloride

INTERVENTIONS:
Drug: aprepitant — 125 mg orally for 7 days
  Other Names: EMEND
  Arms: ARM A
Drug: ondansetron hydrochloride — 24 mg orally for 7 days
  Other Names: Zofran
  Arms: ARM B

SUMMARY:
RATIONALE: Antiemetic drugs, such as aprepitant and ondansetron, may help lessen nausea and vomiting caused by opioids. It is not yet known whether aprepitant is more effective than ondansetron in treating nausea and vomiting caused by opioids in patients with cancer.

PURPOSE: This randomized clinical trial is studying aprepitant to see how well it works compared to ondansetron in treating nausea and vomiting caused by opioids in patients with cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the efficacy of aprepitant as monotherapy for opioid-induced nausea and vomiting (OINV) in comparison to ondansetron hydrochloride in patients who have failed at least one prior anti-emetic agent/regimen.

Secondary

* To determine whether control of OINV improves quality of life.
* To determine if control in OINV decreases pain.
* To determine if control in OINV improves mood.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

* Arm A: Patients receive aprepitant orally once daily for 7 days in the absence of unacceptable toxicity or persistent grade 4 nausea and vomiting.
* Arm B: Patients receive ondansetron hydrochloride orally 3 times daily for 7 days in the absence of unacceptable toxicity or persistent grade 4 nausea and vomiting.

Patients complete the following questionnaires: Functional Assessment of Cancer Therapy-General (FACT-G); Center for Epidemiologic Studies Depression Scale (CES-D); and Brief Pain Index (BPI) at baseline and on day 7. Patients also complete symptom diaries documenting the following: number of episodes (an emetic episode is defined as a simple vomit or retch, or any number of continuous vomits or retches; distinct episodes that are separated by at least 1 minute) of vomiting or retching including the date and time; worst and average degree of nausea (recorded every 2 hours while awake during the first 24 hours after treatment and every 8 hours on days 1-7); and adverse events other than episodes of vomiting and nausea.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* History of malignancy (including hematological malignancies)
* Has pain requiring opioid analgesics
* Nausea and vomiting (associated with opioid analgesic use) that is unrelieved by at least one standard antiemetic regimen (including 5HT3 antagonist and dexamethasone combination therapy)

  * Patients who have failed ondansetron hydrochloride for treatment of opioid-induced nausea and vomiting will be excluded from the study

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Able to assess severity of nausea and vomiting and document it in the diary
* Women must not be pregnant or lactating
* Women of childbearing potential and sexually active males are strongly advised to use an accepted and effective method of contraception
* Urine pregnancy test will be given to women of childbearing age
* No concerns about compliance with medication regimen or medical follow-up (patient must be able to tolerate oral dosing)
* No severe or chronic illness or other causes of nausea and vomiting, that in judgment of the treating physician, will place patient at risk
* No severe gastrointestinal obstruction or active peptic ulcer disease
* Serum ALT and AST < 2 times upper limit of normal (ULN)
* Serum bilirubin < 2 times ULN
* Serum alkaline phosphatase < 2 times ULN

PRIOR CONCURRENT THERAPY:

* No surgery within the past 7 days
* No chemotherapy within the past 7 days
* No total or lower body radiation therapy within the past 7 days
* Patient may not be scheduled to undergo total body irradiation or lower body irradiation, chemotherapy, or surgery during study participation
* Patient must not be taking warfarin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-08; Primary Completion 2008-01 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Control of nausea and vomiting | Day 1 and Day 7

SECONDARY OUTCOMES:
Quality of life | Day 1 and Day 7
Pain control | Day 1 and Day 7
Mood | Day 1 and Day 7
Global satisfaction | Day 1 and Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A. Murphy, MD, Study Chair — Vanderbilt-Ingram Cancer Center